CLINICAL TRIAL: NCT04528303
Title: A Randomized, Controlled Trial of the Effectiveness of Whole Genome Sequencing Versus Whole Exome Sequencing for Screening Patients With Congenital Diarrhea and Enteropathy (CODESeq)
Brief Title: Whole Genome Sequencing Versus Whole Exome Sequencing for Congenital Diarrhea and Enteropahty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: WGS_CODE_01
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Diarrhea, Infantile; Enteropathy
MeSH Terms: conditions — Diarrhea, Infantile; Intestinal Diseases | interventions — Whole Genome Sequencing; Exome Sequencing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole genome sequencing (Experimental)
  Interventions: Genetic: Whole genome sequencing
- Whole exome sequencing (Active Comparator)
  Interventions: Genetic: Whole exome sequencing

INTERVENTIONS:
Genetic: Whole genome sequencing — Genomic sequencing and molecular diagnostic results
  Arms: Whole genome sequencing
Genetic: Whole exome sequencing — Genomic sequencing and molecular diagnostic results
  Arms: Whole exome sequencing

SUMMARY:
This study will seek to determine if whole genome sequencing (WGS) improves diagnostic rates, and outcomes for congenital diarrhea and enteropathy (CODE) patients. The investigator will enroll 180 patients in a randomized controlled study to either WGS or whole exome sequencing (WES). This study is designed to evaluate whether CODE patients would benefit from WGS guided precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic diarrhea lasting greater than 2 months
* Patients with consent from parents or legal guardians
* Biological relative of a patient enrolled in this study.

Exclusion Criteria:

* Chronic diarrhea caused by specific infections, i.e. CMV, Clostridioides difficile
* Chronic diarrhea with necrotizing enterocolitis, short bowel syndrome
* Functional diarrhea
* Patients with previously confirmed monogenic diarrhea
* Patients with poor compliance

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic rates between WGS and WES | Within approximately 60 days of enrollment
  Diagnostic rate of genome and exome based on rate of clinically confirmed diagnoses.

SECONDARY OUTCOMES:
Number of patients receiving precision medicine guided by sequencing results | Within approximately 60 days of enrollment
  Rate of application of precision medicine suggested by the results of WGS or WES.
Mortality of patients | Within approximately 1 year of enrollment
  Mortality of patients after WGS and WES
Rate of parental satisfaction with sequencing | Within one week of patient enrollment
  Parental satisfaction with decision to pursue sequencing based on questionnaire survey
Number of parents who are available for trio sequencing | Within one week of patient enrollment
  Number of subjects in which both parents are available for trio sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, MD,PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Ying Huang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No